CLINICAL TRIAL: NCT02834013
Title: DART: Dual Anti-CTLA-4 and Anti-PD-1 Blockade in Rare Tumors
Brief Title: Nivolumab and Ipilimumab in Treating Patients With Rare Tumors
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2016-01041; NCI-2016-01041 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); S1609 (Other: SWOG); S1609 (Other: CTEP); U10CA180888 (NIH)
Record Dates: First submitted 2016-07-13; First posted 2016-07-15 (Estimated); Last update posted 2026-02-12 (Actual); Status verified 2025-09

CONDITIONS: Acinar Cell Carcinoma; Adenoid Cystic Carcinoma; Adrenal Cortical Carcinoma; Adrenal Gland Pheochromocytoma; Anal Canal Neuroendocrine Carcinoma; Anal Canal Undifferentiated Carcinoma; Angiosarcoma; Apocrine Neoplasm; Appendix Mucinous Adenocarcinoma; Bartholin Gland Transitional Cell Carcinoma; Basal Cell Carcinoma; Bladder Adenocarcinoma; Breast Metaplastic Carcinoma; Cervical Adenocarcinoma; Cholangiocarcinoma; Chordoma; Colorectal Squamous Cell Carcinoma; Desmoid Fibromatosis; Endometrial Transitional Cell Carcinoma; Endometrioid Adenocarcinoma; Esophageal Neuroendocrine Carcinoma; Esophageal Undifferentiated Carcinoma; Extrahepatic Bile Duct Carcinoma; Extramammary Paget Disease; Fallopian Tube Adenocarcinoma; Fallopian Tube Transitional Cell Carcinoma; Fibromyxoid Tumor; Gallbladder Carcinoma; Gastric Neuroendocrine Carcinoma; Gastric Squamous Cell Carcinoma; Gastric Undifferentiated Carcinoma; Gastrointestinal Stromal Tumor; Gestational Trophoblastic Tumor; Giant Cell Carcinoma; Human Papillomavirus-Independent Cervical Adenocarcinoma, Clear Cell-Type; Intestinal Neuroendocrine Carcinoma; Intrahepatic Cholangiocarcinoma; Lung Neuroendocrine Tumor; Lung Sarcomatoid Carcinoma; Major Salivary Gland Carcinoma; Malignant Neoplasm of Unknown Primary; Malignant Odontogenic Neoplasm; Malignant Peripheral Nerve Sheath Tumor; Malignant Solid Neoplasm; Malignant Testicular Sex Cord-Stromal Tumor; Metastatic Pituitary Neuroendocrine Tumor; Minimally Invasive Lung Adenocarcinoma; Mixed Mesodermal (Mullerian) Tumor; Mucinous Adenocarcinoma; Mucinous Cystadenocarcinoma; Nasal Cavity Adenocarcinoma; Nasal Cavity Carcinoma; Nasopharyngeal Carcinoma; Nasopharyngeal Low Grade Papillary Adenocarcinoma; Nasopharyngeal Undifferentiated Carcinoma; Oral Cavity Carcinoma; Oropharyngeal Undifferentiated Carcinoma; Ovarian Adenocarcinoma; Ovarian Germ Cell Tumor; Ovarian Mucinous Adenocarcinoma; Ovarian Squamous Cell Carcinoma; Ovarian Transitional Cell Carcinoma; Pancreatic Acinar Cell Carcinoma; Pancreatic Neuroendocrine Carcinoma; Paraganglioma; Paranasal Sinus Adenocarcinoma; Paranasal Sinus Carcinoma; Parathyroid Gland Carcinoma; PEComa; Penile Squamous Cell Carcinoma; Peritoneal Mesothelial Neoplasm; Placental Choriocarcinoma; Primary Peritoneal High Grade Serous Adenocarcinoma; Pseudomyxoma Peritonei; Rare Disorder; Scrotal Squamous Cell Carcinoma; Seminal Vesicle Adenocarcinoma; Seminoma; Serous Cystadenocarcinoma; Small Intestinal Adenocarcinoma; Small Intestinal Squamous Cell Carcinoma; Spindle Cell Neoplasm; Teratoma With Somatic-Type Malignancy; Testicular Non-Seminomatous Germ Cell Tumor; Thyroid Gland Carcinoma; Tracheal Carcinoma; Transitional Cell Carcinoma; Ureter Adenocarcinoma; Ureter Squamous Cell Carcinoma; Urethral Adenocarcinoma; Urethral Squamous Cell Carcinoma; Vaginal Adenocarcinoma; Vaginal Squamous Cell Carcinoma, Not Otherwise Specified; Vulvar Carcinoma
MeSH Terms: conditions — Carcinoma, Acinar Cell; Carcinoma, Adenoid Cystic; Adrenocortical Carcinoma; Pheochromocytoma; Hemangiosarcoma; Carcinoma, Basal Cell; Cholangiocarcinoma; Chordoma; Desmoid Tumors; Carcinoma, Endometrioid; Bile Duct Neoplasms; Paget Disease, Extramammary; Fibroma; Gallbladder Neoplasms; Gastrointestinal Stromal Tumors; Gestational Trophoblastic Disease; Carcinoma, Giant Cell; Neurofibrosarcoma; Adenocarcinoma, Bronchiolo-Alveolar; Carcinosarcoma; Adenocarcinoma, Mucinous; Cystadenocarcinoma, Mucinous; Nasopharyngeal Carcinoma; Mouth Neoplasms; Somatostatinoma; Paraganglioma; Paranasal Sinus Neoplasms; Parathyroid Neoplasms; Perivascular Epithelioid Cell Neoplasms; Pseudomyxoma Peritonei; Rare Diseases; Seminoma; Cystadenocarcinoma, Serous; Thyroid Neoplasms; Carcinoma, Transitional Cell; Vulvar Neoplasms | interventions — Specimen Handling; Ipilimumab; CTLA-4 Antigen; Magnetic Resonance Spectroscopy; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (nivolumab, ipilimumab) (Experimental): Patients receive nivolumab IV over 30 minutes on days 1, 15, and 29 and ipilimumab IV over 60 minutes on day 1. Treatment repeats every 42 days for up to 17 cycles (2 years) in the absence of disease progression or unacceptable toxicity. Patients who complete 17 cycles (2 years) of therapy, may continue receiving the same treatment with nivolumab and ipilimumab, or receive nivolumab once every 14 or 28 days (2 weeks or 4 weeks) per physician discretion in the absence of disease progression or unacceptable toxicity. Patients who stop treatment prior to the completion of 17 cycles of therapy may receive nivolumab once every 14 or 28 days (2 weeks or 4 weeks) in the absence of disease progression or unacceptable toxicity. Patients undergo ECHO during screening and on study. Patients also undergo MRI or CT throughout the trial. Additionally, patients undergo blood sample collection throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Echocardiography Test; Biological: Ipilimumab; Procedure: Magnetic Resonance Imaging; Biological: Nivolumab
- Arm II (nivolumab) (Experimental): Patients receive nivolumab IV over 30 minutes on days 1, 15 and 29. Treatment repeats every 42 days for up to 17 cycles (2 years) in the absence of disease progression or unacceptable toxicity. After 17 cycles (2 years) of therapy, patients may receive nivolumab once every 14 or 28 days (2 weeks or 4 weeks) in the absence of disease progression or unacceptable toxicity. Patients undergo ECHO during screening and on study. Patients also undergo MRI or CT throughout the trial. Additionally, patients undergo blood sample collection throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Echocardiography Test; Procedure: Magnetic Resonance Imaging; Biological: Nivolumab

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Echocardiography Test — Undergo ECHO
  Other Names: EC; Echocardiography
Biological: Ipilimumab — Given IV
  Other Names: Anti-Cytotoxic T-Lymphocyte-Associated Antigen-4 Monoclonal Antibody; BMS 734016; BMS-734016; BMS734016; Ipilimumab Biosimilar CS1002; MDX 010; MDX-010; MDX-CTLA4; MDX010; Yervoy
  Arms: Arm I (nivolumab, ipilimumab)
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Biological: Nivolumab — Given IV
  Other Names: ABP 206; BCD-263; BMS 936558; BMS-936558; BMS936558; CMAB819; MDX 1106; MDX-1106; MDX1106; NIVO; Nivolumab Biosimilar ABP 206; Nivolumab Biosimilar BCD-263; Nivolumab Biosimilar CMAB819; ONO 4538; ONO-4538; ONO4538; Opdivo

SUMMARY:
This phase II trial studies nivolumab and ipilimumab in treating patients with rare tumors. Immunotherapy with monoclonal antibodies, such as nivolumab and ipilimumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread.

This trial enrolls participants for the following cohorts based on condition:

1. Epithelial tumors of nasal cavity, sinuses, nasopharynx: A) Squamous cell carcinoma with variants of nasal cavity, sinuses, and nasopharynx and trachea (excluding laryngeal, nasopharyngeal cancer [NPC], and squamous cell carcinoma of the head and neck [SCCHN]) B) Adenocarcinoma and variants of nasal cavity, sinuses, and nasopharynx (closed to accrual 07/27/2018)
2. Epithelial tumors of major salivary glands (closed to accrual 03/20/2018)
3. Salivary gland type tumors of head and neck, lip, esophagus, stomach, trachea and lung, breast and other location (closed to accrual)
4. Undifferentiated carcinoma of gastrointestinal (GI) tract
5. Adenocarcinoma with variants of small intestine (closed to accrual 05/10/2018)
6. Squamous cell carcinoma with variants of GI tract (stomach small intestine, colon, rectum, pancreas) (closed to accrual 10/17/2018)
7. Fibromixoma and low grade mucinous adenocarcinoma (pseudomixoma peritonei) of the appendix and ovary (closed to accrual 03/20/2018)
8. Rare pancreatic tumors including acinar cell carcinoma, mucinous cystadenocarcinoma or serous cystadenocarcinoma. Pancreatic adenocarcinoma is not eligible (closed to accrual)
9. Intrahepatic cholangiocarcinoma (closed to accrual 03/20/2018)
10. Extrahepatic cholangiocarcinoma and bile duct tumors (closed to accrual 03/20/2018)
11. Sarcomatoid carcinoma of lung
12. Bronchoalveolar carcinoma lung. This condition is now also referred to as adenocarcinoma in situ, minimally invasive adenocarcinoma, lepidic predominant adenocarcinoma, or invasive mucinous adenocarcinoma
13. Non-epithelial tumors of the ovary: A) Germ cell tumor of ovary B) Mullerian mixed tumor and adenosarcoma (closed to accrual 03/30/2018)
14. Trophoblastic tumor: A) Choriocarcinoma (closed to accrual)
15. Transitional cell carcinoma other than that of the renal, pelvis, ureter, or bladder (closed to accrual)
16. Cell tumor of the testes and extragonadal germ tumors: A) Seminoma and testicular sex cord cancer B) Non seminomatous tumor C) Teratoma with malignant transformation (closed to accrual)
17. Epithelial tumors of penis - squamous adenocarcinoma cell carcinoma with variants of penis (closed to accrual)
18. Squamous cell carcinoma variants of the genitourinary (GU) system
19. Spindle cell carcinoma of kidney, pelvis, ureter
20. Adenocarcinoma with variants of GU system (excluding prostate cancer) (closed to accrual 07/27/2018)
21. Odontogenic malignant tumors
22. Pancreatic neuroendocrine tumor (PNET) (formerly named: Endocrine carcinoma of pancreas and digestive tract.) (closed to accrual)
23. Neuroendocrine carcinoma including carcinoid of the lung (closed to accrual 12/19/2017)
24. Pheochromocytoma, malignant (closed to accrual)
25. Paraganglioma (closed to accrual 11/29/2018)
26. Carcinomas of pituitary gland, thyroid gland parathyroid gland and adrenal cortex (closed to accrual)
27. Desmoid tumors
28. Peripheral nerve sheath tumors and NF1-related tumors (closed to accrual 09/19/2018)
29. Malignant giant cell tumors
30. Chordoma (closed to accrual 11/29/2018)
31. Adrenal cortical tumors (closed to accrual 06/27/2018)
32. Tumor of unknown primary (Cancer of Unknown Primary; CuP) (closed to accrual 12/22/2017)
33. Not Otherwise Categorized (NOC) Rare Tumors [To obtain permission to enroll in the NOC cohort, contact: S1609SC@swog.org] (closed to accrual 03/15/2019)
34. Adenoid cystic carcinoma (closed to accrual 02/06/2018)
35. Vulvar cancer (closed to accrual)
36. MetaPLASTIC carcinoma (of the breast) (closed to accrual)
37. Gastrointestinal stromal tumor (GIST) (closed to accrual 09/26/2018)
38. Perivascular epithelioid cell tumor (PEComa)
39. Apocrine tumors/extramammary Paget's disease (closed to accrual)
40. Peritoneal mesothelioma
41. Basal cell carcinoma (temporarily closed to accrual 04/29/2020)
42. Clear cell cervical cancer
43. Esthenioneuroblastoma (closed to accrual)
44. Endometrial carcinosarcoma (malignant mixed Mullerian tumors) (closed to accrual)
45. Clear cell endometrial cancer
46. Clear cell ovarian cancer (closed to accrual)
47. Gestational trophoblastic disease (GTD)
48. Gallbladder cancer
49. Small cell carcinoma of the ovary, hypercalcemic type
50. PD-L1 amplified tumors
51. Angiosarcoma
52. High-grade neuroendocrine carcinoma (pancreatic neuroendocrine tumor [PNET] should be enrolled in Cohort 22; prostatic neuroendocrine carcinomas should be enrolled into Cohort 53). Small cell lung cancer is not eligible (closed to accrual)
53. Treatment-emergent small-cell neuroendocrine prostate cancer (t-SCNC)

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1 overall response rate (ORR) in subsets of patients with advanced rare cancers treated with ipilimumab plus nivolumab combination immunotherapy.

II. To evaluate the overall response rate (ORR) in patients with gestational trophoblastic tumors treated with ipilimumab plus nivolumab combination immunotherapy.

III. To evaluate the RECIST v1.1 overall response rate (ORR) in patients PD-L1 amplified cancers treated with nivolumab immunotherapy.

SECONDARY OBJECTIVES:

I. To evaluate toxicities in each cohort. II. To estimate overall survival (OS), progression-free survival (PFS), clinical benefit rate; and to estimate immune related (i)RECIST ORR (iORR), and iRECIST PFS (iPFS) across cohorts and within each cohort.

OUTLINE: Patients are assigned to 1 of 2 arms.

ARM I (ALL COHORTS EXCEPT THE PD-L1 AMPLIFIED COHORT): Patients receive nivolumab intravenously (IV) over 30 minutes on days 1, 15, and 29 and ipilimumab IV over 60 minutes on day 1. Treatment repeats every 42 days for up to 17 cycles (2 years) in the absence of disease progression or unacceptable toxicity. Patients who complete 17 cycles (2 years) of therapy, may continue receiving the same treatment with nivolumab and ipilimumab, or receive nivolumab once every 14 or 28 days (2 weeks or 4 weeks) per physician discretion in the absence of disease progression or unacceptable toxicity. Patients who stop treatment prior to the completion of 17 cycles of therapy may receive nivolumab once every 14 or 28 days (2 weeks or 4 weeks) in the absence of disease progression or unacceptable toxicity. Patients undergo echocardiography (ECHO) during screening and on study. Patients also undergo magnetic resonance imaging (MRI) or computed tomography (CT) throughout the trial. Additionally, patients undergo blood sample collection throughout the trial.

ARM II (PD-L1 AMPLIFIED COHORT): Patients receive nivolumab IV over 30 minutes on days 1, 15 and 29. Treatment repeats every 42 days for up to 17 cycles (2 years) in the absence of disease progression or unacceptable toxicity. After 17 cycles (2 years) of therapy, patients may receive nivolumab once every 14 or 28 days (2 weeks or 4 weeks) in the absence of disease progression or unacceptable toxicity. Patients undergo ECHO during screening and on study. Patients also undergo MRI or CT throughout the trial. Additionally, patients undergo blood sample collection throughout the trial.

After completion of study treatment, patients are followed up for 10 years from registration.

ELIGIBILITY:
Inclusion Criteria:

* Patients are eligible under ONE of the following criteria:

  * For all cohorts except the gestational trophoblastic disease (GTD) (Cohort #47), patients must have histologically and/or biochemically confirmed rare cancer and must be able to submit specimens; to be eligible for the GTD cohort: patients must have disease confirmed by quantitative serum beta-human chorionic gonadotropin (hCG) within 28 days prior to registration and must be able to submit blood specimens (tissue submission is not required for patients who will be registered to the GTD cohort [Cohort #47]); NOTE: Subsequent to site's Institutional Review Board (IRB) approval of revision 3, patients are NOT required to participate in EAY131 "National Cancer Institute (NCI)-Molecular Analysis for Therapy Choice (MATCH)" to register to S1609 OR
  * FOR PATIENTS WITH PD-L1 AMPLIFICATION (COHORT #50) ONLY: All solid tumors (excluding lymphoma) are allowed for the PD-L1 amplified cohort if they have PD-L1 amplification; patients may be considered for registration to the PD-L1 amplified cohort (Cohort #50) with the confirmation of at least one of the study chairs; PD-L1 amplification is defined as having deoxyribonucleic acid (DNA) copy number of equal to or greater than six by any of the following Clinical Laboratory Improvement Act (CLIA)-approved lab; (Immunohisochemistry [IHC] and fluorescence in situ hybridization [FISH] are not allowed); the assay must be done at or after the diagnosis of advanced disease, but PRIOR TO REGISTRATION; NOTE: patients with PD-L1 overexpression by IHC or PD-L1 amplification by FISH do not quality for this cohort; OR
  * FOR PATIENTS ENROLLED IN EAY131 "NCI-MATCH" PRIOR TO EAY131 ADDENDUM 10 ONLY: Patients must have histologically confirmed rare cancer that did not have a match to a molecularly-guided therapy on EAY131 "NCI-MATCH" protocol or who are off protocol treatment on EAY131, "NCI-MATCH" and have no further molecularly-matched treatment recommendations per EAY131, "NCI-MATCH" or who are otherwise unable to receive EAY131, "NCI-MATCH" therapy
* Patients who do not qualify for one of the histologic cohorts and are not on the ineligible histology list may be considered for registration in the "Not Otherwise Categorized" Rare Tumors cohort with confirmation of at least one of the study chairs via email

  * NOTE: The "Not Otherwise Categorized" Rare Tumors cohort was permanently closed to accrual on 3/15/2019
* Patients who are determined to have a rare cancer with unknown primary site are eligible under cohort #32 (tumor of unknown primary [cancer of unknown primary; CuP]), provided that there is histologic documentation of metastatic malignancy with no discernible primary site identified from histopathologic review, physical exam and associated cross-sectional imaging of the chest, abdomen, and pelvis

  * NOTE: The "Tumor of unknown primary (Cancer of Unknown Primary; CuP" cohort was permanently closed to accrual on 12/22/2017
* Patients must also meet one of the following:

  * Patients must have progressed following at least one line of standard systemic therapy and there must not be other approved/standard therapy available that has been shown to prolong overall survival (i.e. in a randomized trial against another standard treatment or by comparison to historical controls); patients who cannot receive other standard therapy that has been shown to prolonged survival due to medical issues will be eligible, if other eligibility criteria are met; OR
  * Patients for whose disease no standard treatment exists that has been shown to prolong overall survival
* For all cohorts except the GTD cohort (Cohort #47): Patients must have a diagnostic quality computed tomography (CT) scan or magnetic resonance imaging (MRI), performed within 28 days prior to registration, which demonstrates measurable disease, as defined in RECIST v. 1.1; scans must include imaging of the chest, abdomen and pelvis, with the exception of patients with head/neck cancer, who must have imaging of the chest, abdomen, pelvis and neck; if there is clinical suspicion for bone metastases at the time of enrollment (in the judgement of the treating investigator) bone scan should be performed; bone scans done within 42 days prior to registration may be used to establish baseline condition at registration
* No other prior malignancy is allowed except for the following:

  * Adequately managed stage I or II cancer from which the patient is currently in complete remission
  * Any other cancer from which the patient has been disease free for one year
  * Adequately managed stage I or II follicular thyroid or prostate cancer is also eligible, wherein patient is not required to be in complete remission
  * Note: Second primary tumors are not allowed concurrent with any of the eligible rare cancers
* For all cohorts except the PD-L1 amplified tumors cohort (Cohort # 50): Patients may have received either prior anti-CTLA4 or other prior anti-PD-1/anti-PD-L1 therapy, but not both, provided that it is completed >= 4 weeks prior to registration. To be eligible for the PD-L1 amplified tumors cohort (Cohort #50): Patients must not have received anti-PD-1/anti-PD-L1 therapy; prior anti-CTLA-4 is allowed provided that it is completed >= 4 weeks prior to registration
* Patients who had prior grade 3 or higher immune-related adverse event (e.g. pneumonitis, hepatitis, colitis, endocrinopathy) with prior immunotherapy (e.g. cancer vaccine, cytokine, etc.) are not eligible
* Patients with clinically controlled thyroiditis or pituitary disorders on stable replacement therapy are eligible
* Patients are not eligible if they have had or are planned for solid organ transplant
* Patients with autoimmune disease who are otherwise eligible must not have received steroid and immunosuppressive therapy within 28 days prior to registration
* Patients with brain metastases or primary brain tumors must have completed treatment, surgery or radiation therapy >= 28 days prior to registration and have stable disease at time of registration; these patients must also have a CT or MRI of the brain to evaluate for CNS disease within 42 days prior to registration to S1609; metastatic brain parenchymal disease must have been treated and patient must be off steroids for 7 days prior to registration
* Patients must not currently be receiving any other investigational agents or any other systemic anti-cancer therapy (including radiation, excluding RANKL inhibitors and bisphosphonates); in event patient recently received any other systemic anti-cancer therapy, patient must be off therapy at least 7 days prior to registration and any therapy-induced toxicity must have recovered to =< grade 1, except alopecia and =< grade 2 neuropathy which are allowed; any planned radiation therapy must be completed before registration to S1609
* Patients must not have prior history of allergy or known hypersensitivity to nivolumab or ipilimumab
* Hormonal or endocrine blockade is permitted as long as patient has demonstrated progression on prior therapy (e.g. gonadotrophin releasing hormone [GnRH], somatostatin); long-acting somatostatin analogs (including octreotide) and androgen deprivation treatment (including long-acting leuprolide) are permitted while on protocol therapy
* Patients must be >= 18 years of age
* Patients must have a Zubrod performance status of 0-2
* Absolute neutrophil count (ANC) >= 1,000/mcL (within 28 days prior to registration)
* Platelets >= 75,000/mcL (within 28 days prior to registration)
* Hemoglobin >= 8 g/dL (within 28 days prior to registration)
* Total bilirubin =< 2.0 x institutional upper limit of normal (IULN) or for documented/suspected Gilbert's disease, total bilirubin =< 3.0 x IULN (within 28 days prior to registration)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) both =< 3 x IULN (within 28 days prior to registration)
* Serum creatinine =< 2.0 x IULN (within 28 days prior to registration)
* Creatinine clearance (CrCl) >= 50 mL/min., as estimated by the Cockcroft and Gault formula; estimated creatinine clearance is based on actual body weight (within 28 days prior to registration)
* Patients must have adequate thyroid function, as evidenced by either thyroid-stimulating hormone (TSH) or, free thyroxine (T4) serum tests demonstrating values within the normal range, within 28 days prior to registration; at pre-registration, if TSH is not within normal limits, then free T4 must be performed and must be within normal range for patient to be eligible; Note: TSH, with reflex T4 (if TSH is abnormal) is allowable if per institutional standard, provided that free T4 is within normal range; patients who have undergone thyroidectomy or who are on thyroid suppression for their cancer are not required to have normal TSH and free T4
* Patients must have adequate adrenal axis function, as evidenced by cortisol levels within institutional normal ranges (ante meridiem [AM] cortisol preferred), OR adrenocorticotropic hormone (ACTH) values within the institutional normal ranges within 28 days prior to registration; if cortisol levels are not within normal limits prior to registration, then ACTH must be performed and must be within normal ranges for patient to be eligible; Note: Neither cortisol nor ACTH levels are required for patients with primary adrenal tumors (e.g. adrenocortical carcinoma)
* For women of childbearing potential, the local investigator must rule out pregnancy; Except for Cohorts 13 and 47, where tumor types may express beta-hCG, women of childbearing potential must have a serum or urine pregnancy test within 7 days prior to registration; for Cohorts 13 and 47, where tumor types may produce hCG (e.g. germ cell tumors or trophoblastic disease), other pregnancy exclusion methods should be used to rule out pregnancy, such as ultrasound examination, documented history of effective contraception, or documented infertility; all females of childbearing potential must have been demonstrated not to be pregnant within 7 days prior to registration and agree to use birth control throughout study and for 23 weeks after completion of protocol therapy; patients must not be pregnant or nursing due to risk of fetal or nursing infant harm; women of childbearing potential must have agreed to use an effective contraceptive method; a woman is considered to be of "childbearing potential" if she has had menses at any time in the preceding 12 consecutive months; in addition to routine contraceptive methods, "effective contraception" also includes heterosexual celibacy and surgery intended to prevent pregnancy (or with a side-effect of pregnancy prevention) defined as a hysterectomy, bilateral oophorectomy or bilateral tubal ligation; however, if at any point a previously celibate patient chooses to become heterosexually active during the time period for use of contraceptive measures outlined in the protocol, she is responsible for beginning contraceptive measures
* Men of reproductive potential must have agreed to use birth control throughout the study and for 31 weeks after completion of protocol therapy; in addition to routine contraceptive methods, "effective contraception" also includes heterosexual celibacy and surgery intended to prevent pregnancy (vasectomy); however, if at any point a previously celibate patient chooses to become heterosexually active during the time period for use of contraceptive measures outlined in the protocol, he is responsible for beginning contraceptive measures
* Patients must not have known active hepatitis B virus (HBV) or hepatitis virus (HCV) infection at time of registration; patients with HBV or HCV that have an undetectable viral load and no residual hepatic impairment are eligible
* Patients who are known to be human immunodeficiency virus (HIV)-positive at registration are eligible at the time of registration:

  * CD4+ cell count greater or equal to 250 cells/mm^3
  * No history of non-malignancy acquired immunodeficiency syndrome (AIDS)-defining conditions other than historical low CD4+ cell counts
* Patients must not have active autoimmune disease that has required systemic treatment in past 2 years (i.e., with use of disease modifying agents, immunosuppressive drugs, or corticosteroids with prednisone dose >= 10 mg); replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment; autoimmune diseases include but are not limited to autoimmune hepatitis, inflammatory bowel disease (including ulcerative colitis and Crohn's disease), as well as symptomatic disease (e.g.: rheumatoid arthritis, systemic progressive sclerosis [scleroderma], systemic lupus erythematosus, autoimmune vasculitis [e.g., Wegener's granulomatosis]); central nervous system (CNS) or motor neuropathy considered of autoimmune origin (e.g., Guillain-Barre syndrome and Myasthenia gravis, multiple sclerosis or glomerulonephritis); vitiligo, alopecia, hypothyroidism on stable doses of thyroid replacement therapy, psoriasis not requiring systemic therapy within the past 2 years is permitted; short-term steroid premedication for contrast allergy is permitted
* Patients must not have any uncontrolled intercurrent illness including (not limited to): symptomatic congestive heart failure (CHF) (New York Heart Association [NYHA] III/IV), unstable angina pectoris or coronary angioplasty, or stenting within 24 weeks prior to registration, unstable cardiac arrhythmia (ongoing cardiac dysrhythmias of NCI Common Terminology Criteria for Adverse Events [CTCAE] version [v] 4 grade >= 2), known psychiatric illness that would limit study compliance, intra-cardiac defibrillators, known cardiac metastases, or abnormal cardiac valve morphology (>= grade 3)

  * Note: Patients with history of CHF or patients who are deemed at risk because of underlying cardiovascular disease or exposure to cardiotoxic drugs should have an electrocardiogram (EKG) and echocardiogram (ECHO), as clinically indicated, at baseline and at the start of each cycle; patients who have evidence at baseline (or subsequently) of CHF, myocardial infarction (MI), cardiomyopathy, or myositis cardiac evaluation (NYHA I/II) should have additional consult by a cardiologist, including review of EKG, creatine phosphokinase (CPK), troponin, echocardiogram, as clinically indicated
* Patients must have amylase or lipase within =< 1.5 x IULN without symptoms of pancreatitis at registration, within 28 days prior to registration
* Patients must not have symptomatic interstitial lung disease or pneumonitis
* Patients must have fully recovered from any adverse effects of major surgery (to =< grade 1) at least 14 days prior to registration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 818 (Estimated)
Dates: Start 2017-01-30 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | Up to 10 years
  Defined as confirmed and unconfirmed complete and partial response. Assessed by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.

SECONDARY OUTCOMES:
Incidence of adverse events | Up to 10 years
  Graded by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. Assuming 16 eligible patients per stratum, this will be sufficient to estimate each binary version of this endpoint within +/- 25% (95% confidence interval).
Best response | Up to 10 years
  Calculated from the sequence of RECIST 1.1 and immune-related (i)RECIST objectives. Assuming 16 eligible patients per stratum, this will be sufficient to estimate each binary version of this endpoint within +/- 25% (95% confidence interval).
Clinical benefit rate | 6 months
  Defined as complete response, partial response, or stable disease, estimated using both RECIST and iRECIST. Assuming 16 eligible patients per stratum, this will be sufficient to estimate each binary version of this endpoint within +/- 25% (95% confidence interval).
Overall survival (OS) | From date of registration to date of death due to any cause, assessed up to 10 years
  Estimated using both RECIST and immune-related (ir) RESIST criteria (RC). Assuming 16 eligible patients per stratum, this will be sufficient to estimate each binary version of this endpoint within +/- 25% (95% confidence interval).
Progression free survival (PFS) | From date of registration to date of first documentation of progression or symptomatic deterioration or death, assessed up to 10 years
  Estimated using both RECIST and irRC. Assuming 16 eligible patients per stratum, this will be sufficient to estimate each binary version of this endpoint within +/- 25% (95% confidence interval).

CONTACTS AND LOCATIONS:
Overall Officials: Sandip P Patel, Principal Investigator — SWOG Cancer Research Network
Locations (1009):
- United States (1008):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - University of South Alabama Mitchell Cancer Institute, Mobile, Alabama
  - Anchorage Associates in Radiation Medicine, Anchorage, Alaska
  - Anchorage Radiation Therapy Center, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Fairbanks Memorial Hospital, Fairbanks, Alaska
  - CTCA at Western Regional Medical Center, Goodyear, Arizona
  - Kingman Regional Medical Center, Kingman, Arizona
  - Cancer Center at Saint Joseph's, Phoenix, Arizona
  - Highlands Oncology Group - Fayetteville, Fayetteville, Arkansas
  - Mercy Hospital Fort Smith, Fort Smith, Arkansas
  - CHI Saint Vincent Cancer Center Hot Springs, Hot Springs, Arkansas
  - NEA Baptist Memorial Hospital and Fowler Family Cancer Center - Jonesboro, Jonesboro, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Highlands Oncology Group - Rogers, Rogers, Arkansas
  - Highlands Oncology Group, Springdale, Arkansas
  - Kaiser Permanente-Anaheim, Anaheim, California
  - Kaiser Permanente-Deer Valley Medical Center, Antioch, California
  - Mission Hope Medical Oncology - Arroyo Grande, Arroyo Grande, California
  - PCR Oncology, Arroyo Grande, California
  - Sutter Auburn Faith Hospital, Auburn, California
  - Sutter Cancer Centers Radiation Oncology Services-Auburn, Auburn, California
  - AIS Cancer Center at San Joaquin Community Hospital, Bakersfield, California
  - Kaiser Permanente-Baldwin Park, Baldwin Park, California
  - Kaiser Permanente-Bellflower, Bellflower, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Keck Medicine of USC Buena Park, Buena Park, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Mills-Peninsula Medical Center, Burlingame, California
  - Sutter Cancer Centers Radiation Oncology Services-Cameron Park, Cameron Park, California
  - Mercy Cancer Center - Carmichael, Carmichael, California
  - Mercy San Juan Medical Center, Carmichael, California
  - Eden Hospital Medical Center, Castro Valley, California
  - UC Irvine Health Cancer Center-Newport, Costa Mesa, California
  - Sutter Davis Hospital, Davis, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Epic Care-Dublin, Dublin, California
  - Kaiser Permanente Dublin, Dublin, California
  - Mercy Cancer Center - Elk Grove, Elk Grove, California
  - Bay Area Breast Surgeons Inc, Emeryville, California
  - Epic Care Partners in Cancer Care, Emeryville, California
  - Kaiser Permanente-Fontana, Fontana, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Palo Alto Medical Foundation-Fremont, Fremont, California
  - Kaiser Permanente-Fresno, Fresno, California
  - Kaiser Permanente South Bay, Harbor City, California
  - Keck Medicine of USC Huntington Beach, Huntington Beach, California
  - Kaiser Permanente-Irvine, Irvine, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Keck Medicine of USC Koreatown, Los Angeles, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Kaiser Permanente West Los Angeles, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Contra Costa Regional Medical Center, Martinez, California
  - Fremont - Rideout Cancer Center, Marysville, California
  - Mercy Cancer Center, Merced, California
  - Memorial Medical Center, Modesto, California
  - Kaiser Permanente-Modesto, Modesto, California
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - Palo Alto Medical Foundation-Gynecologic Oncology, Mountain View, California
  - Providence Queen of The Valley, Napa, California
  - USC Norris Oncology/Hematology-Newport Beach, Newport Beach, California
  - Sutter Cancer Research Consortium, Novato, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Bay Area Tumor Institute, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Kaiser Permanente-Ontario, Ontario, California
  - Saint Joseph Hospital - Orange, Orange, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Desert Regional Medical Center, Palm Springs, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Kaiser Permanente - Panorama City, Panorama City, California
  - Keck Medical Center of USC Pasadena, Pasadena, California
  - Eisenhower Medical Center, Rancho Mirage, California
  - Kaiser Permanente- Marshall Medical Offices, Redwood City, California
  - Kaiser Permanente-Redwood City, Redwood City, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Kaiser Permanente-Riverside, Riverside, California
  - Mercy Cancer Center - Rocklin, Rocklin, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - Sutter Roseville Medical Center, Roseville, California
  - Kaiser Permanente Downtown Commons, Sacramento, California
  - Mercy Cancer Center - Sacramento, Sacramento, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - Kaiser Permanente Sacramento Medical Center, Sacramento, California
  - UC San Diego Medical Center - Hillcrest, San Diego, California
  - Kaiser Permanente-San Diego Mission, San Diego, California
  - Kaiser Permanente-San Diego Zion, San Diego, California
  - Sharp Memorial Hospital, San Diego, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Pacific Central Coast Health Center-San Luis Obispo, San Luis Obispo, California
  - Kaiser Permanente-San Marcos, San Marcos, California
  - Mills Health Center, San Mateo, California
  - Kaiser Permanente-San Rafael, San Rafael, California
  - Kaiser San Rafael-Gallinas, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Palo Alto Medical Foundation-Santa Cruz, Santa Cruz, California
  - Mission Hope Medical Oncology - Santa Maria, Santa Maria, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Providence Medical Foundation - Santa Rosa, Santa Rosa, California
  - Sutter Pacific Medical Foundation, Santa Rosa, California
  - Providence Santa Rosa Memorial Hospital, Santa Rosa, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - Gene Upshaw Memorial Tahoe Forest Cancer Center, Truckee, California
  - Kaiser Permanente Medical Center-Vacaville, Vacaville, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Epic Care Cyberknife Center, Walnut Creek, California
  - Woodland Memorial Hospital, Woodland, California
  - Kaiser Permanente-Woodland Hills, Woodland Hills, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - The Medical Center of Aurora, Aurora, Colorado
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Boulder Community Foothills Hospital, Boulder, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Rocky Mountain Cancer Centers - Centennial, Centennial, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - UCHealth Memorial Hospital Central, Colorado Springs, Colorado
  - Memorial Hospital North, Colorado Springs, Colorado
  - Saint Francis Cancer Center, Colorado Springs, Colorado
  - Cancer Center of Colorado at Sloan's Lake, Denver, Colorado
  - Denver Health Medical Center, Denver, Colorado
  - Kaiser Permanente-Franklin, Denver, Colorado
  - National Jewish Health-Main Campus, Denver, Colorado
  - The Women's Imaging Center, Denver, Colorado
  - AdventHealth Porter, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - Saint Joseph Hospital - Cancer Centers of Colorado, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - CommonSpirit Cancer Center Mercy, Durango, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Mountain Blue Cancer Care Center - Swedish, Englewood, Colorado
  - Rocky Mountain Cancer Centers - Swedish, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - The Melanoma and Skin Cancer Institute, Englewood, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Valley View Hospital Cancer Center, Glenwood Springs, Colorado
  - Mountain Blue Cancer Care Center, Golden, Colorado
  - National Jewish Health-Western Hematology Oncology, Golden, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - Grand Valley Oncology, Grand Junction, Colorado
  - Banner North Colorado Medical Center, Greeley, Colorado
  - Rocky Mountain Cancer Centers-Greenwood Village, Greenwood Village, Colorado
  - Good Samaritan Hospital - Cancer Centers of Colorado, Lafayette, Colorado
  - Kaiser Permanente-Rock Creek, Lafayette, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - AdventHealth Littleton, Littleton, Colorado
  - Kaiser Permanente-Lone Tree, Lone Tree, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - Banner North Colorado Medical Center - Loveland Campus, Loveland, Colorado
  - AdventHealth Parker, Parker, Colorado
  - Rocky Mountain Cancer Centers-Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Rocky Mountain Cancer Centers - Pueblo, Pueblo, Colorado
  - National Jewish Health-Northern Hematology Oncology, Thornton, Colorado
  - Rocky Mountain Cancer Centers-Thornton, Thornton, Colorado
  - Intermountain Health Lutheran Hospital, Wheat Ridge, Colorado
  - Smilow Cancer Hospital-Derby Care Center, Derby, Connecticut
  - Smilow Cancer Hospital Care Center-Fairfield, Fairfield, Connecticut
  - Smilow Cancer Hospital Care Center - Guilford, Guilford, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Smilow Cancer Center/Yale-New Haven Hospital, New Haven, Connecticut
  - Yale University, New Haven, Connecticut
  - Yale-New Haven Hospital North Haven Medical Center, North Haven, Connecticut
  - Stamford Hospital/Bennett Cancer Center, Stamford, Connecticut
  - Smilow Cancer Hospital Care Center-Trumbull, Trumbull, Connecticut
  - Smilow Cancer Hospital-Waterbury Care Center, Waterbury, Connecticut
  - Veterans Affairs Connecticut Healthcare System-West Haven Campus, West Haven, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Beebe South Coastal Health Campus, Millville, Delaware
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - TidalHealth Nanticoke / Allen Cancer Center, Seaford, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - AdventHealth Altamonte, Altamonte Springs, Florida
  - Mount Sinai Comprehensive Cancer Center at Aventura, Aventura, Florida
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - AdventHealth Kissimmee, Kissimmee, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - AdventHealth Medical Group Urology at Orlando, Orlando, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - AdventHealth East Orlando, Orlando, Florida
  - Memorial Hospital West, Pembroke Pines, Florida
  - Moffitt Cancer Center-International Plaza, Tampa, Florida
  - Moffitt Cancer Center - McKinley Campus, Tampa, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - AdventHealth Winter Park, Winter Park, Florida
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Piedmont Hospital, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - John B Amos Cancer Center, Columbus, Georgia
  - Atlanta VA Medical Center, Decatur, Georgia
  - Piedmont Fayette Hospital, Fayetteville, Georgia
  - Harbin Clinic Medical Oncology and Clinical Research, Rome, Georgia
  - Low Country Cancer Care, Savannah, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Summit Cancer Care-Candler, Savannah, Georgia
  - South Georgia Medical Center/Pearlman Cancer Center, Valdosta, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Island Urology, Honolulu, Hawaii
  - Queen's Cancer Cenrer - POB I, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hawaii Cancer Care Inc-Liliha, Honolulu, Hawaii
  - Hawaii Diagnostic Radiology Services LLC, Honolulu, Hawaii
  - Kuakini Medical Center, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Straub Medical Center - Kahului Clinic, Kahului, Hawaii
  - Castle Medical Center, Kailua, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Hawaii Cancer Care - Westridge, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Queen's Cancer Center - Pearlridge, ‘Aiea, Hawaii
  - Straub Pearlridge Clinic, ‘Aiea, Hawaii
  - The Cancer Center of Hawaii-Pali Momi, ‘Aiea, Hawaii
  - The Queen's Medical Center - West Oahu, ‘Ewa Beach, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Walter Knox Memorial Hospital, Emmett, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - OSF Saint Anthony's Health Center, Alton, Illinois
  - Rush-Copley Medical Center, Aurora, Illinois
  - OSF Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Loyola Center for Health at Burr Ridge, Burr Ridge, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Mount Sinai Hospital Medical Center, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - Rush MD Anderson Cancer Center, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Loyola Medicine Homer Glen, Homer Glen, Illinois
  - Presence Saint Mary's Hospital, Kankakee, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Marjorie Weinberg Cancer Center at Loyola-Gottlieb, Melrose Park, Illinois
  - SSM Health Good Samaritan, Mount Vernon, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - University of Chicago Medicine-Orland Park, Orland Park, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Southwest Illinois Health Services LLP, Swansea, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Midwestern Regional Medical Center, Zion, Illinois
  - IU Health West Hospital, Avon, Indiana
  - IU Health North Hospital, Carmel, Indiana
  - Deaconess Clinic Downtown, Evansville, Indiana
  - Parkview Regional Medical Center, Fort Wayne, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Sidney and Lois Eskenazi Hospital, Indianapolis, Indiana
  - Springmill Medical Center, Indianapolis, Indiana
  - Memorial Regional Cancer Center Day Road, Mishawaka, Indiana
  - Chancellor Center for Oncology, Newburgh, Indiana
  - Reid Health, Richmond, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - McFarland Clinic - Boone, Boone, Iowa
  - Saint Anthony Regional Hospital, Carroll, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Alegent Health Mercy Hospital, Council Bluffs, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - Broadlawns Medical Center, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - McFarland Clinic - Trinity Cancer Center, Fort Dodge, Iowa
  - UI Healthcare Mission Cancer and Blood - Fort Dodge, Fort Dodge, Iowa
  - McFarland Clinic - Jefferson, Jefferson, Iowa
  - McFarland Clinic - Marshalltown, Marshalltown, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Coffeyville Regional Medical Center, Coffeyville, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - University of Kansas Clinical Research Center, Fairway, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Central Care Cancer Center - Garden City, Garden City, Kansas
  - Saint Catherine Hospital, Garden City, Kansas
  - Central Care Cancer Center - Great Bend, Great Bend, Kansas
  - HaysMed, Hays, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - University of Kansas Cancer Center-West, Kansas City, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas-Manhattan, Manhattan, Kansas
  - Cancer Center of Kansas - McPherson, McPherson, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - The University of Kansas Cancer Center - Olathe, Olathe, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - University of Kansas Hospital-Indian Creek Campus, Overland Park, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Freeman Physician Group of Pittsburg, Pittsburg, Kansas
  - Mercy Hospital Pittsburg, Pittsburg, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Commonwealth Cancer Center-Corbin, Corbin, Kentucky
  - Saint Joseph Hospital, Lexington, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - Saint Joseph London, London, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - Saints Mary and Elizabeth Hospital, Louisville, Kentucky
  - UofL Health Medical Center Northeast, Louisville, Kentucky
  - Saint Joseph Mount Sterling, Mount Sterling, Kentucky
  - Jewish Hospital Medical Center South, Shepherdsville, Kentucky
  - Baton Rouge General Medical Center, Baton Rouge, Louisiana
  - Hematology/Oncology Clinic PLLC, Baton Rouge, Louisiana
  - Ochsner Health Center-Summa, Baton Rouge, Louisiana
  - Medical Center of Baton Rouge, Baton Rouge, Louisiana
  - Ochsner High Grove, Baton Rouge, Louisiana
  - Ochsner Medical Center Kenner, Kenner, Louisiana
  - East Jefferson General Hospital, Metairie, Louisiana
  - LSU Healthcare Network / Metairie Multi-Specialty Clinic, Metairie, Louisiana
  - Louisiana State University Health Science Center, New Orleans, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Lafayette Family Cancer Center-EMMC, Brewer, Maine
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - UPMC Western Maryland, Cumberland, Maryland
  - Frederick Memorial Hospital, Frederick, Maryland
  - FMH James M Stockman Cancer Institute, Frederick, Maryland
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Lahey Medical Center-Peabody, Peabody, Massachusetts
  - Mercy Medical Center, Springfield, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - Hickman Cancer Center, Adrian, Michigan
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - University of Michigan Rogel Cancer Center, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health Medical Center - Brighton, Brighton, Michigan
  - University of Michigan - Brighton Center for Specialty Care, Brighton, Michigan
  - Henry Ford Cancer Institute-Downriver, Brownstown, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health Medical Center - Canton, Canton, Michigan
  - Caro Cancer Center, Caro, Michigan
  - Chelsea Hospital, Chelsea, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Hematology Oncology Consultants-Clarkston, Clarkston, Michigan
  - Newland Medical Associates-Clarkston, Clarkston, Michigan
  - Henry Ford Hematology Oncology - Hayes, Clinton Township, Michigan
  - Henry Ford Macomb Hospital-Clinton Township, Clinton Township, Michigan
  - Corewell Health Dearborn Hospital, Dearborn, Michigan
  - Henry Ford Medical Center-Fairlane, Dearborn, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - Henry Ford River District Hospital, East China Township, Michigan
  - OSF Saint Francis Hospital and Medical Group, Escanaba, Michigan
  - Cancer Hematology Centers - Flint, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Henry Ford Saint John Hospital - Academic, Grosse Pointe Woods, Michigan
  - Henry Ford Saint John Hospital - Breast, Grosse Pointe Woods, Michigan
  - Henry Ford Saint John Hospital - Van Elslander, Grosse Pointe Woods, Michigan
  - Allegiance Health, Jackson, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Beacon Kalamazoo Cancer Center, Kalamazoo, Michigan
  - Beacon Kalamazoo, Kalamazoo, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Hope Cancer Clinic, Livonia, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Henry Ford Saint John Hospital - Macomb Medical, Macomb, Michigan
  - Henry Ford Warren Hospital - Breast Macomb, Macomb, Michigan
  - Schoolcraft Memorial Hospital, Manistique, Michigan
  - Saint Mary's Oncology/Hematology Associates of Marlette, Marlette, Michigan
  - Monroe Cancer Center, Monroe, Michigan
  - Toledo Clinic Cancer Centers-Monroe, Monroe, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Corewell Health Lakeland Hospitals - Niles Hospital, Niles, Michigan
  - Cancer and Hematology Centers of Western Michigan - Norton Shores, Norton Shores, Michigan
  - Henry Ford Health Providence Novi Hospital, Novi, Michigan
  - Henry Ford Medical Center-Columbus, Novi, Michigan
  - Hope Cancer Center, Pontiac, Michigan
  - Michigan Healthcare Professionals Pontiac, Pontiac, Michigan
  - Newland Medical Associates-Pontiac, Pontiac, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Huron Medical Center PC, Port Huron, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - Corewell Health Reed City Hospital, Reed City, Michigan
  - Henry Ford Rochester Hospital, Rochester Hills, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Corewell Health Lakeland Hospitals - Saint Joseph Hospital, Saint Joseph, Michigan
  - Henry Ford Macomb Health Center - Shelby Township, Shelby, Michigan
  - Henry Ford Health Providence Southfield Hospital, Southfield, Michigan
  - Bhadresh Nayak MD PC-Sterling Heights, Sterling Heights, Michigan
  - MyMichigan Medical Center Tawas, Tawas City, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Advanced Breast Care Center PLLC, Warren, Michigan
  - Henry Ford Health Warren Hospital, Warren, Michigan
  - Henry Ford Madison Heights Hospital - Breast, Warren, Michigan
  - Henry Ford Warren Hospital - GLCMS, Warren, Michigan
  - Macomb Hematology Oncology PC, Warren, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - Saint Mary's Oncology/Hematology Associates of West Branch, West Branch, Michigan
  - Henry Ford Wyandotte Hospital, Wyandotte, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Huron Gastroenterology PC, Ypsilanti, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Riverwood Healthcare Center, Aitkin, Minnesota
  - Essentia Health - Baxter Clinic, Baxter, Minnesota
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Minnesota Oncology - Burnsville, Burnsville, Minnesota
  - Cambridge Medical Center, Cambridge, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Saint Mary's - Detroit Lakes Clinic, Detroit Lakes, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Essentia Health - Ely Clinic, Ely, Minnesota
  - Lake Region Healthcare Corporation-Cancer Care, Fergus Falls, Minnesota
  - Essentia Health - Fosston, Fosston, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Essentia Health - International Falls Clinic, International Falls, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - Essentia Health - Moose Lake Clinic, Moose Lake, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - Essentia Health - Park Rapids, Park Rapids, Minnesota
  - Fairview Northland Medical Center, Princeton, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Sanford Thief River Falls Medical Center, Thief River Falls, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Sanford Cancer Center Worthington, Worthington, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - Baptist Memorial Hospital and Cancer Center-Golden Triangle, Columbus, Mississippi
  - Baptist Cancer Center-Grenada, Grenada, Mississippi
  - Gulfport Memorial Hospital, Gulfport, Mississippi
  - Hattiesburg Clinic - Hematology/Oncology Clinic, Hattiesburg, Mississippi
  - Forrest General Hospital / Cancer Center, Hattiesburg, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Union County, New Albany, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Oxford, Oxford, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Desoto, Southhaven, Mississippi
  - Mercy Oncology and Hematology - Clayton-Clarkson, Ballwin, Missouri
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Mercy Cancer Center - Cape Girardeau, Cape Girardeau, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Saint Luke's Hospital, Chesterfield, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - MU Health Care Goldschmidt Cancer Center, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - University Health Truman Medical Center, Kansas City, Missouri
  - Kansas City Veterans Affairs Medical Center, Kansas City, Missouri
  - The University of Kansas Cancer Center-South, Kansas City, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Phelps Health Delbert Day Cancer Institute, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Mercy Infusion Center - Chippewa, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Mercy Hospital Washington, Washington, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Saint Vincent Frontier Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Nebraska Cancer Specialists/Oncology Hematology West PC, Grand Island, Nebraska
  - Fred and Pamela Buffett Cancer Center - Kearney, Kearney, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Saint Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Nebraska Cancer Specialists/Oncology Hematology West PC - MECC, Omaha, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Oncology Associates PC, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Hematology and Oncology Consultants PC, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Midlands Community Hospital, Papillion, Nebraska
  - Carson Tahoe Regional Medical Center, Carson City, Nevada
  - Cancer and Blood Specialists-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Horizon Ridge, Henderson, Nevada
  - Las Vegas Cancer Center-Henderson, Henderson, Nevada
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - Las Vegas Urology - Green Valley, Henderson, Nevada
  - Las Vegas Urology - Pebble, Henderson, Nevada
  - Oncology Las Vegas - Henderson, Henderson, Nevada
  - Urology Specialists of Nevada - Green Valley, Henderson, Nevada
  - Las Vegas Urology - Pecos, Las Vegas, Nevada
  - Desert West Surgery, Las Vegas, Nevada
  - OptumCare Cancer Care at Charleston, Las Vegas, Nevada
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Hope Cancer Care of Nevada, Las Vegas, Nevada
  - Cancer and Blood Specialists-Shadow, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - Urology Specialists of Nevada - Central, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Maryland Parkway, Las Vegas, Nevada
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-San Martin, Las Vegas, Nevada
  - Las Vegas Prostate Cancer Center, Las Vegas, Nevada
  - Las Vegas Urology - Sunset, Las Vegas, Nevada
  - Urology Specialists of Nevada - Southwest, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - Cancer Therapy and Integrative Medicine, Las Vegas, Nevada
  - Ann M Wierman MD LTD, Las Vegas, Nevada
  - Cancer and Blood Specialists-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Tenaya, Las Vegas, Nevada
  - Las Vegas Urology - Cathedral Rock, Las Vegas, Nevada
  - Las Vegas Urology - Smoke Ranch, Las Vegas, Nevada
  - Oncology Las Vegas - Tenaya, Las Vegas, Nevada
  - OptumCare Cancer Care at MountainView, Las Vegas, Nevada
  - Urology Specialists of Nevada - Northwest, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Town Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Las Vegas Cancer Center-Medical Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Centennial Hills, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - University Cancer Center, Las Vegas, Nevada
  - Hope Cancer Care of Nevada-Pahrump, Pahrump, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Saint Mary's Regional Medical Center, Reno, Nevada
  - Radiation Oncology Associates, Reno, Nevada
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Dartmouth Cancer Center - Manchester, Manchester, New Hampshire
  - Dartmouth Cancer Center - Nashua, Nashua, New Hampshire
  - Morristown Medical Center, Morristown, New Jersey
  - Chilton Medical Center, Pompton, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - Inspira Medical Center Vineland, Vineland, New Jersey
  - Lovelace Medical Center-Saint Joseph Square, Albuquerque, New Mexico
  - Southwest Gynecologic Oncology Associates Inc, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - New Mexico Oncology Hematology Consultants, Albuquerque, New Mexico
  - Presbyterian Kaseman Hospital, Albuquerque, New Mexico
  - Memorial Medical Center-Las Cruces, Las Cruces, New Mexico
  - Presbyterian Rust Medical Center/Jorgensen Cancer Center, Rio Rancho, New Mexico
  - Christus Saint Vincent Regional Cancer Center, Santa Fe, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - Arnot Ogden Medical Center/Falck Cancer Center, Elmira, New York
  - Glens Falls Hospital, Glens Falls, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - University of Rochester, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - AdventHealth Infusion Center Asheville, Asheville, North Carolina
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - AdventHealth Infusion Center Haywood, Clyde, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - AdventHealth Hendersonville, Hendersonville, North Carolina
  - Onslow Memorial Hospital, Jacksonville, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - ECU Health Oncology Kenansville, Kenansville, North Carolina
  - ECU Health Oncology Kinston, Kinston, North Carolina
  - ECU Health Oncology Richlands, Richlands, North Carolina
  - AdventHealth Infusion Center Weaverville, Weaverville, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Essentia Health Cancer Center-South University Clinic, Fargo, North Dakota
  - Sanford South University Medical Center, Fargo, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Essentia Health - Jamestown Clinic, Jamestown, North Dakota
  - Indu and Raj Soin Medical Center, Beavercreek, Ohio
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Saint Elizabeth Boardman Hospital, Boardman, Ohio
  - Cleveland Clinic Mercy Hospital, Canton, Ohio
  - Dayton Physicians LLC-Miami Valley South, Centerville, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Kenwood, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - TriHealth Cancer Institute-Anderson, Cincinnati, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Mount Carmel East Hospital, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Dayton Physician LLC - Englewood, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Delaware Radiation Oncology, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Columbus Oncology and Hematology Associates, Dublin, Ohio
  - Dublin Methodist Hospital, Dublin, Ohio
  - Armes Family Cancer Center, Findlay, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Orion Cancer Care, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Dayton Physicians LLC-Atrium, Franklin, Ohio
  - Dayton Physicians LLC-Wayne, Greenville, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Mount Carmel Grove City Hospital, Grove City, Ohio
  - Zangmeister Center Grove City, Grove City, Ohio
  - Greater Dayton Cancer Center, Kettering, Ohio
  - First Dayton Cancer Care, Kettering, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Saint Rita's Medical Center, Lima, Ohio
  - OhioHealth Mansfield Hospital, Mansfield, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - OhioHealth Marion General Hospital, Marion, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - Toledo Radiation Oncology at Northwest Ohio Onocolgy Center, Maumee, Ohio
  - Dayton Physicians LLC-Signal Point, Middletown, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Mount Carmel New Albany Surgical Hospital, New Albany, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - Mercy Health - Perrysburg Hospital, Perrysburg, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - Dayton Physicians LLC-Wilson, Sidney, Ohio
  - Springfield Regional Cancer Center, Springfield, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - Mercy Health - Saint Vincent Hospital, Toledo, Ohio
  - Mercy Health - Saint Anne Hospital, Toledo, Ohio
  - Mercy Health Sylvania Radiation Oncology Center, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Dayton Physicians LLC - Troy, Troy, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Saint Joseph Warren Hospital, Warren, Ohio
  - South Pointe Hospital, Warrensville Heights, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Saint Elizabeth Youngstown Hospital, Youngstown, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - Cancer Centers of Southwest Oklahoma Research, Lawton, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Cancer Treatment Centers of America, Tulsa, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Saint Alphonsus Cancer Care Center-Baker City, Baker City, Oregon
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Kaiser Sunnyside Medical Center, Clackamas, Oregon
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Saint Alphonsus Cancer Care Center-Ontario, Ontario, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Kaiser Permanente Northwest, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Saint Charles Health System-Redmond, Redmond, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - UPMC-Heritage Valley Health System Beaver, Beaver, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Christiana Care Health System-Concord Health Center, Chadds Ford, Pennsylvania
  - UPMC Hillman Cancer Center - Passavant - Cranberry, Cranberry Township, Pennsylvania
  - Doylestown Hospital, Doylestown, Pennsylvania
  - Pocono Medical Center, East Stroudsburg, Pennsylvania
  - Saint Vincent Hospital, Erie, Pennsylvania
  - UPMC Cancer Centers - Arnold Palmer Pavilion, Greensburg, Pennsylvania
  - Lehigh Valley Hospital-Hazleton, Hazleton, Pennsylvania
  - IRMC Cancer Center, Indiana, Pennsylvania
  - Jefferson Hospital, Jefferson Hills, Pennsylvania
  - UPMC-Johnstown/John P. Murtha Regional Cancer Center, Johnstown, Pennsylvania
  - UPMC Cancer Center at UPMC McKeesport, McKeesport, Pennsylvania
  - Forbes Hospital, Monroeville, Pennsylvania
  - UPMC Hillman Cancer Center - Monroeville, Monroeville, Pennsylvania
  - UPMC Hillman Cancer Center in Coraopolis, Moon Township, Pennsylvania
  - UPMC Hillman Cancer Center - Part of Frick Hospital, Mount Pleasant, Pennsylvania
  - Arnold Palmer Cancer Center Medical Oncology Norwin, N. Huntingdon, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Eastern Regional Medical Center, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - UPMC-Magee Womens Hospital, Pittsburgh, Pennsylvania
  - UPMC-Presbyterian Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Margaret, Pittsburgh, Pennsylvania
  - West Penn Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - UPMC-Shadyside Hospital, Pittsburgh, Pennsylvania
  - UPMC-Passavant Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Clair Hospital Cancer Center, Pittsburgh, Pennsylvania
  - Pottstown Hospital, Pottstown, Pennsylvania
  - UPMC Cancer Center at UPMC Northwest, Seneca, Pennsylvania
  - UPMC Uniontown Hospital Radiation Oncology, Uniontown, Pennsylvania
  - UPMC Cancer Center-Washington, Washington, Pennsylvania
  - UPMC Washington Hospital Radiation Oncology, Washington, Pennsylvania
  - UPMC West Mifflin-Cancer Center Jefferson, West Mifflin, Pennsylvania
  - Wexford Health and Wellness Pavilion, Wexford, Pennsylvania
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Cancer Institute - Laurens, Clinton, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Gibbs Cancer Center-Gaffney, Gaffney, South Carolina
  - Tidelands Georgetown Memorial Hospital, Georgetown, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - North Grove Medical Park, Spartanburg, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Spartanburg Medical Center - Mary Black Campus, Spartanburg, South Carolina
  - SMC Center for Hematology Oncology Union, Union, South Carolina
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Memorial Hospital, Chattanooga, Tennessee
  - Baptist Memorial Hospital and Cancer Center-Collierville, Collierville, Tennessee
  - Vanderbilt-Ingram Cancer Center Cool Springs, Franklin, Tennessee
  - Pulmonary Medicine Center of Chattanooga-Hixson, Hixson, Tennessee
  - Baptist Memorial Hospital and Cancer Center-Memphis, Memphis, Tennessee
  - Vanderbilt Breast Center at One Hundred Oaks, Nashville, Tennessee
  - Meharry Medical College, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Memorial GYN Plus, Ooltewah, Tennessee
  - Saint Joseph Regional Cancer Center, Bryan, Texas
  - Parkland Memorial Hospital, Dallas, Texas
  - Baylor University Medical Center, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Fort Worth, Fort Worth, Texas
  - Lyndon Baines Johnson General Hospital, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - UT Southwestern Clinical Center at Richardson/Plano, Richardson, Texas
  - University Hospital, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - American Fork Hospital / Huntsman Intermountain Cancer Center, American Fork, Utah
  - Sandra L Maxwell Cancer Center, Cedar City, Utah
  - Farmington Health Center, Farmington, Utah
  - Logan Regional Hospital, Logan, Utah
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - Riverton Hospital, Riverton, Utah
  - Utah Cancer Specialists-Salt Lake City, Salt Lake City, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - South Jordan Health Center, South Jordan, Utah
  - Saint George Regional Medical Center, St. George, Utah
  - Central Vermont Medical Center/National Life Cancer Treatment, Berlin Corners, Vermont
  - University of Vermont Medical Center, Burlington, Vermont
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - Dartmouth Cancer Center - North, Saint Johnsbury, Vermont
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - Cancer Care Center at Island Hospital, Anacortes, Washington
  - MultiCare Auburn Medical Center, Auburn, Washington
  - Virginia Mason Bainbridge Island Medical Center, Bainbridge Island, Washington
  - Overlake Medical Center, Bellevue, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Saint Elizabeth Hospital, Enumclaw, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Virginia Mason Federal Way Medical Center, Federal Way, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - Tacoma/Valley Radiation Oncology Centers-Gig Harbor, Gig Harbor, Washington
  - MultiCare Gig Harbor Medical Park, Gig Harbor, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Northwest Cancer Clinic, Kennewick, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Virginia Mason Lynnwood Medical Center, Lynnwood, Washington
  - Skagit Regional Health Cancer Care Center, Mount Vernon, Washington
  - Skagit Valley Hospital, Mount Vernon, Washington
  - Jefferson Healthcare, Port Townsend, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - Peninsula Cancer Center, Poulsbo, Washington
  - MultiCare Good Samaritan Hospital, Puyallup, Washington
  - Tacoma/Valley Radiation Oncology Centers-Puyallup, Puyallup, Washington
  - Valley Medical Center, Renton, Washington
  - Virginia Mason Medical Center, Seattle, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - Kaiser Permanente Washington, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - University of Washington Medical Center - Montlake, Seattle, Washington
  - PeaceHealth United General Medical Center, Sedro-Woolley, Washington
  - Providence Regional Cancer System-Shelton, Shelton, Washington
  - Saint Michael Cancer Center, Silverdale, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - Downtown, Spokane, Washington
  - Spokane Valley Cancer Center-Mayfair, Spokane, Washington
  - Spokane Valley Cancer Center-Mission, Spokane, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - North, Spokane, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - Valley, Spokane Valley, Washington
  - Tacoma/Valley Radiation Oncology Centers-Jackson Hall, Tacoma, Washington
  - Franciscan Research Center-Northwest Medical Plaza, Tacoma, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - MultiCare Tacoma General Hospital, Tacoma, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington
  - Tacoma/Valley Radiation Oncology Centers-Saint Joe's, Tacoma, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Legacy Cancer Institute Medical Oncology and Day Treatment, Vancouver, Washington
  - Legacy Salmon Creek Hospital, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - Wenatchee Valley Hospital and Clinics, Wenatchee, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - Providence Regional Cancer System-Yelm, Yelm, Washington
  - Edwards Comprehensive Cancer Center, Huntington, West Virginia
  - Ascension Saint Elizabeth Hospital, Appleton, Wisconsin
  - Duluth Clinic Ashland, Ashland, Wisconsin
  - Northwest Wisconsin Cancer Center, Ashland, Wisconsin
  - Ascension Southeast Wisconsin Hospital - Elmbrook Campus, Brookfield, Wisconsin
  - Ascension Calumet Hospital, Chilton, Wisconsin
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - Marshfield Clinic Cancer Center at Sacred Heart, Eau Claire, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Ascension Saint Francis - Reiman Cancer Center, Franklin, Wisconsin
  - Ascension Southeast Wisconsin Hospital - Franklin, Franklin, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Marshfield Medical Center - Ladysmith, Ladysmith, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Saint Vincent Hospital Cancer Center at Marinette, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Ascension Columbia Saint Mary's Hospital Ozaukee, Mequon, Wisconsin
  - Ascension Southeast Wisconsin Hospital - Saint Joseph Campus, Milwaukee, Wisconsin
  - Ascension Columbia Saint Mary's Hospital - Milwaukee, Milwaukee, Wisconsin
  - Ascension Saint Francis Hospital, Milwaukee, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - Ascension Mercy Hospital, Oshkosh, Wisconsin
  - Ascension All Saints Hospital, Racine, Wisconsin
  - Aspirus Cancer Care - James Beck Cancer Center, Rhinelander, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - HSHS Saint Nicholas Hospital, Sheboygan, Wisconsin
  - Aspirus Cancer Care - Stevens Point, Stevens Point, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Ascension Medical Group Southeast Wisconsin - Mayfair Road, Wauwatosa, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Cheyenne Regional Medical Center-West, Cheyenne, Wyoming
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming
- FHP Health Center-Guam, Tamuning, Guam

REFERENCES:
- [Derived] Patel SP, Fisher J, Chae YK, Soto LS, Kasi A, Konda B, Walshauser M, Parra E, Zhang J, Duault C, Gonzalez-Kozlova E, Manyam G, Zhang J, Chen H, Duose DY, Laberiano Fernandez C, Luthra R, Al-Atrash G, Kim-Schulze S, Maecker HT, Wistuba II, Gnjatic S, Lee JJ, Zhang J, Magner CM, Chen HX, Sharon E, Othus M, Ryan CW, Blanke C, Haymaker CL, Kurzrock R. Phase II basket trial of Dual Anti-CTLA-4 and anti-PD-1 blockade in Rare Tumors (DART) SWOG S1609: pancreatic neuroendocrine neoplasm (PNEN) cohort. J Immunother Cancer. 2025 Jun 30;13(6):e011760. doi: 10.1136/jitc-2025-011760. PMID 40588371
- [Derived] Patel SP, Cano-Linson E, Chae YK, Schokrpur S, Lao CD, Powers BC, Victor AI, Onitilo AA, Shin S, Takebe N, Threlkel S, McLeod CM, Chen HX, Sharon E, Othus M, Ryan CW, Blanke CD, Kurzrock R. Dual anti-CTLA-4 and anti-PD-1 blockade in metastatic basal cell carcinoma. NPJ Precis Oncol. 2025 Jan 24;9(1):24. doi: 10.1038/s41698-024-00798-1. PMID 39856213
- [Derived] Chae YK, Othus M, Patel SP, Gerber DE, Tanvetyanon T, Kim HS, Chung LI, McLeod CM, Lopez G, Chen HX, Sharon E, Streicher H, Ryan CW, Blanke CD, Kurzrock R. Phase II trial of dual anti-CTLA-4 and anti-PD-1 blockade in rare tumors SWOG/NCI experience: invasive mucinous or non-mucinous lepidic adenocarcinoma of the lung (formerly bronchioloalveolar carcinoma). Ther Adv Med Oncol. 2024 Nov 22;16:17588359241293401. doi: 10.1177/17588359241293401. eCollection 2024. PMID 39583952
- [Derived] Chae YK, Othus M, Patel S, Powers B, Hsueh CT, Govindarajan R, Bucur S, Kim HS, Chung LI, McLeod C, Chen HX, Sharon E, Streicher H, Ryan CW, Blanke C, Kurzrock R. Phase II basket trial of dual anti-CTLA-4 and anti-PD-1 blockade in rare tumors (DART) SWOG S1609: the desmoid tumors. J Immunother Cancer. 2024 Sep 28;12(9):e009128. doi: 10.1136/jitc-2024-009128. PMID 39343510
- [Derived] Patel SP, Othus M, Chae YK, Huynh T, Tan B, Kuzel T, McLeod C, Lopez G, Chen HX, Sharon E, Streicher H, Ryan CW, Blanke C, Kurzrock R. Phase II basket trial of Dual Anti-CTLA-4 and Anti-PD-1 blockade in Rare Tumors (DART) SWOG S1609: adrenocortical carcinoma cohort. J Immunother Cancer. 2024 Jul 27;12(7):e009074. doi: 10.1136/jitc-2024-009074. PMID 39067873
- [Derived] Patel SP, Guadarrama E, Chae YK, Dennis MJ, Powers BC, Liao CY, Ferri WA Jr, George TJ, Sharon E, Ryan CW, Othus M, Lopez G, Blanke CD, Kurzrock R. SWOG 1609 cohort 48: anti-CTLA-4 and anti-PD-1 for advanced gallbladder cancer. Cancer. 2024 Sep 1;130(17):2918-2927. doi: 10.1002/cncr.35243. Epub 2024 Feb 15. PMID 38358334
- [Derived] Adams S, Othus M, Patel SP, Miller KD, Chugh R, Schuetze SM, Chamberlin MD, Haley BJ, Storniolo AMV, Reddy MP, Anderson SA, Zimmerman CT, O'Dea AP, Mirshahidi HR, Ahnert JR, Brescia FJ, Hahn O, Raymond JM, Biggs DD, Connolly RM, Sharon E, Korde LA, Gray RJ, Mayerson E, Plets M, Blanke CD, Chae YK, Kurzrock R. A Multicenter Phase II Trial of Ipilimumab and Nivolumab in Unresectable or Metastatic Metaplastic Breast Cancer: Cohort 36 of Dual Anti-CTLA-4 and Anti-PD-1 Blockade in Rare Tumors (DART, SWOG S1609). Clin Cancer Res. 2022 Jan 15;28(2):271-278. doi: 10.1158/1078-0432.CCR-21-2182. Epub 2021 Oct 29. PMID 34716198
- [Derived] Wagner MJ, Othus M, Patel SP, Ryan C, Sangal A, Powers B, Budd GT, Victor AI, Hsueh CT, Chugh R, Nair S, Leu KM, Agulnik M, Sharon E, Mayerson E, Plets M, Blanke C, Streicher H, Chae YK, Kurzrock R. Multicenter phase II trial (SWOG S1609, cohort 51) of ipilimumab and nivolumab in metastatic or unresectable angiosarcoma: a substudy of dual anti-CTLA-4 and anti-PD-1 blockade in rare tumors (DART). J Immunother Cancer. 2021 Aug;9(8):e002990. doi: 10.1136/jitc-2021-002990. PMID 34380663
- [Derived] Patel SP, Mayerson E, Chae YK, Strosberg J, Wang J, Konda B, Hayward J, McLeod CM, Chen HX, Sharon E, Othus M, Ryan CW, Plets M, Blanke CD, Kurzrock R. A phase II basket trial of Dual Anti-CTLA-4 and Anti-PD-1 Blockade in Rare Tumors (DART) SWOG S1609: High-grade neuroendocrine neoplasm cohort. Cancer. 2021 Sep 1;127(17):3194-3201. doi: 10.1002/cncr.33591. Epub 2021 Apr 21. PMID 33882143
- [Derived] Dai C, Liang S, Sun B, Kang J. The Progress of Immunotherapy in Refractory Pituitary Adenomas and Pituitary Carcinomas. Front Endocrinol (Lausanne). 2020 Dec 11;11:608422. doi: 10.3389/fendo.2020.608422. eCollection 2020. PMID 33362722
- [Derived] Patel SP, Othus M, Chae YK, Giles FJ, Hansel DE, Singh PP, Fontaine A, Shah MH, Kasi A, Baghdadi TA, Matrana M, Gatalica Z, Korn WM, Hayward J, McLeod C, Chen HX, Sharon E, Mayerson E, Ryan CW, Plets M, Blanke CD, Kurzrock R. A Phase II Basket Trial of Dual Anti-CTLA-4 and Anti-PD-1 Blockade in Rare Tumors (DART SWOG 1609) in Patients with Nonpancreatic Neuroendocrine Tumors. Clin Cancer Res. 2020 May 15;26(10):2290-2296. doi: 10.1158/1078-0432.CCR-19-3356. Epub 2020 Jan 22. PMID 31969335